CLINICAL TRIAL: NCT05964634
Title: Effect of Peripapillary Atrophy Based on Optical Coherence Tomography to Diagnose Primary Open Angle Glaucoma in High Myopia
Brief Title: Effect of Peripapillary Atrophy to Diagnose Glaucoma in High Myopia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yiqing Li, associate research fellow, Zhongshan Ophthalmic Center, Sun Yat-sen University
Other Study IDs: 2023KYPJ105
Record Dates: First submitted 2023-05-11; First posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Myopia; Refractive Errors; Eye Diseases; Glaucoma, Primary Open Angle; Peripapillary Atrophy
Keywords: high myopia; glaucoma; Peripapillary Atrophy; Optical Coherence Tomography
MeSH Terms: conditions — Myopia; Refractive Errors; Eye Diseases; Glaucoma, Open-Angle; Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- myopic glaucoma: Patiens who have high myopia with primary open angle glaucoma
  Interventions: Diagnostic Test: OCT imaging
- healthy myopia: Patiens who have high myopia without primary open angle glaucoma
  Interventions: Diagnostic Test: OCT imaging

INTERVENTIONS:
Diagnostic Test: OCT imaging — Image J or Spectralis OCT built-in software package was used to manually locate and measure the area and width of the temporal parapapillary atrophy.

SUMMARY:
This study intends to analyze the characteristics between peripapillary retinal nerve fiber layer thickness and peripapillary area in high myopia with or without glaucoma

DETAILED DESCRIPTION:
Glaucoma is the leading cause of irreversible blindness in the world. Myopia is a risk factor for glaucoma. With the rising prevalence of both myopia and glaucoma in an ageing population, the occurrence of these two ocular conditions in the same patient is likely to increase. It was estimated that there were 163 million people who have high myopia in 2000, and the population with high myopia would increase to almost one billion (9.8% of the world population) worldwide by 2050.

There is often a diagnostic challenge to the clinician, since the detection of glaucomatous optic nerve damage in highly myopic eyes is difficult. Recently, the subclassification of peripapillary area could potentially be used to differentiate myopic eyes with and without glaucoma according to OCT findings.

However, the characteristics of peripapillary atrophy have not been fully applied in the diagnosis of high myopia and glaucoma.

In view of the above problems, the purpose of this study is to analyze the peripapillary area based on optical coherence tomography and it may be a specific marker for identifying high myopia with primary open angle glaucoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Equivalent spherical ≤-6D or axial length ≥26.5mm.
3. High myopia with primary open angle glaucoma, such as anterior chamber angle is opening, optic rim defect, RNFL loss, etc.
4. The peripapillary region can be accurately defined Based on OCT.

Exclusion Criteria:

(1) Exclusion criteria for high myopia group:

1. History of glaucoma and elevated intraocular pressure.
2. History of uveitis or intraocular surgery.
3. History of other retinal optic nerve or related systemic diseases.
4. The examination results are unreliable, such as poor image quality.

(2) Exclusion criteria for high myopia with primary open angle glaucoma group:

1. Others nervous system diseases, such as visual field loss or optic nerve damage.
2. Others non-glaucomatous ocular pathologies may affect the visual field or retinal nerve fiber layer status, such as retinal diseases, uveitis, or ocular surgery history.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have high myopia with or without glaucoma.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of circumpapillary retinal nerve fiber layer thickness changes within 12 months | 1 years
  The circle with a diameter of 3.46 mm is scanned by Spectralis OCT instrument with the optic disc as the center and the RNFL thickness was calculated by built-in software.
Evaluation of the area of the peripapillary area changes within 12 months | 1 year
  The results of Spectralis OCT instrument are exported, and used Image J or Spectralis OCT built-in software package to manually locate and measure the area of the temporal parapapillary area
Evaluation of the width of the peripapillary area changes within 12 months | 1 year
  The results of Spectralis OCT instrument are exported, and used Image J or Spectralis OCT built-in software package to manually locate and measure the width of the temporal parapapillary area

SECONDARY OUTCOMES:
Demographic characteristics | 1 day of enrollment
  Including but not limited to gender, age, duration of illness
blood pressure | 1 day of enrollment
  Demographic characteristics
BMI | 1 day of enrollment
  weight (lb) / [height (in)]2
Best corrected visual acuity | 1 day of enrollment
  Best corrected visual acuity after refractive error correction using the ETDRS chart
Evaluation of the intraocular pressure changes within 12 mouths | 1 year
  IOP is measured by goldmann tonometer.
Evaluation of the visual field changes within 12 mouths | 1 year
  Assess the degree of visual function damage
Axial length | 1 day of enrollment
  axial length is measured using A-type ultrasound.
Evaluation of the fundus changes within 12 months | 1 year
  Fundus photography uses kowa fundus camera
Ocular anterior segment structure | 1 day of enrollment
  The ocular anterior segment structure uses lit-lamp biomicroscope

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dai Y, Jonas JB, Huang H, Wang M, Sun X. Microstructure of parapapillary atrophy: beta zone and gamma zone. Invest Ophthalmol Vis Sci. 2013 Mar 19;54(3):2013-8. doi: 10.1167/iovs.12-11255. PMID 23462744
- [Background] Wang YX, Panda-Jonas S, Jonas JB. Optic nerve head anatomy in myopia and glaucoma, including parapapillary zones alpha, beta, gamma and delta: Histology and clinical features. Prog Retin Eye Res. 2021 Jul;83:100933. doi: 10.1016/j.preteyeres.2020.100933. Epub 2020 Dec 9. PMID 33309588
- See also: beta zone and gamma zone defined based on OCT — https://pubmed.ncbi.nlm.nih.gov/23462744/
- See also: Microstructure of parapapillary atrophy — https://pubmed.ncbi.nlm.nih.gov/33309588/